CLINICAL TRIAL: NCT05915247
Title: Phase I, Randomised, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Subcutaneous Single Ascending Doses of HER-096 to Healthy Volunteer Subjects
Brief Title: Single Ascending Doses of HER-096 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herantis Pharma Plc. (Industry)
Collaborators: Clinical Research Services Turku - CRST Oy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-XC-CL; 2022-003283-24 (EudraCT Number)
Record Dates: First submitted 2023-05-08; First posted 2023-06-22 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Part 1: single ascending doses of up to six dosing cohorts Part 2: single dose defined based on the Part 1 data
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Part 1) (Placebo Comparator): Corresponding volumes of placebo solution according to the dosing cohort administered as a s.c. injection.
  Interventions: Drug: Placebo
- HER-096 (Part 1) (Active Comparator): Single ascending doses of HER-096 up to six dosing cohorts administered as a s.c. injection.
  Interventions: Drug: HER-096
- HER-096 (Part 2) (Active Comparator): A single dose of HER-096 will be administered as a s.c. injection.
  Interventions: Drug: HER-096

INTERVENTIONS:
Drug: HER-096 — Administered as a single dose via s.c. injection
  Arms: HER-096 (Part 1); HER-096 (Part 2)
Drug: Placebo — Administered as a single dose via s.c. injection
  Other Names: 0.9% physiological saline; Sodium chloride 9 mg/ml
  Arms: Placebo (Part 1)

SUMMARY:
This study evaluates the safety and tolerability of HER-096 in healthy volunteer subjects by comparing the effects of active study treatment HER-096 to placebo (0.9% physiological saline). In addition, the pharmacokinetic profile of HER-096 in humans will be investigated. The investigational medicinal products will be administered as a single dose by subcutaneous injection.

DETAILED DESCRIPTION:
This is a Phase I, double-blind, placebo-controlled, clinical study, in which safety, tolerability and pharmacokinetic profile of HER-096 will be investigated after a subcutaneously (s.c.) administered single ascending doses of HER-096 to healthy volunteer subjects (HVS).

Altogether 60-64 HVS will be enrolled into the study and the study will be conducted in two parts, part 1 being randomised and part 2 being open-label. In part 1, up to 48 young male HVS will be randomised 6:2 either to receive HER-096 or placebo (0.9% physiological saline) solution. In part 1, up to 6 dosing cohorts have been planned with single ascending doses of HER-096. In part 2, 12-16 older and elderly HVS, both males and females, will be administered with single dose of HER-096 to evaluate the blood-brain-barrier penetration of HER-096. The investigational medicinal products (HER-096 or placebo solution) will be administered as a s.c. injection.

The total duration of the study will be up to 36 days for each subject, consisting of screening and treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and written informed consent and alert and oriented to person, place, time and situation at the time of the informed consent.
2. Sufficient command of the Finnish language.
3. Age 20-45 years for Part 1 and 50-75 years for Part 2.
4. Male sex for Part 1, and male or female for Part 2.
5. Body mass index (BMI) 18-30 kg/m2.
6. Good general health.

Exclusion Criteria:

1. Predicted poor compliance with study procedures, restrictions and requirements.
2. Veins unsuitable for repeated venipuncture or cannulation.
3. History or evidence of current clinically significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, haematological, metabolic-endocrine, neurological, urogenital or psychiatric disorder. Subjects with any type of generalized seizures in adulthood must be excluded. Personal or first-degree family history of congenital long QT syndrome or sudden death of a first-degree relative suspected to be due to long QT syndrome will also exclude the subject.
4. History of any type of cancer, except for the age group of >50 years, where a history of successfully treated cancer may be allowed.
5. Susceptibility to severe allergic reactions, e.g. history of anaphylactic shock.
6. Any condition requiring regular concomitant medication (including non-prescriptional over-the-counter drugs), or likely to need any concomitant medication during the study.
7. Use of any medication that might affect the study results or cause a health risk for the subject within 2 weeks prior to IMP administration.
8. Any clinically significant abnormalities in screening laboratory test results, vital signs or physical examination findings that might influence the results of the study or cause a health risk for the subject if he/she takes part in the study.
9. Coagulopathy, thrombocytopenia, use of anticoagulants or other antithrombotic agents.
10. Positive serology to human immunodeficiency virus antibodies (HIVAgAb), hepatitis C virus antibodies (HCVAb) or hepatitis B surface antigen (HBsAg).
11. Any clinically significant 12-lead ECG abnormality.
12. HR < 45 bpm or > 85 bpm, systolic blood pressure (BP) < 90 mmHg or > 150 mmHg, or diastolic BP < 50 mmHg or > 90 mmHg.
13. History of alcohol or drug abuse within the last 5 years, or current regular use of illicit drugs or excessive use of alcohol.
14. Positive breath test for alcohol or positive urine screening test result for drugs of abuse.
15. Current use of nicotine-containing products of more than 5 cigarettes or equivalent per day, or inability to refrain from using nicotine-containing products.
16. Inability to refrain from consuming caffeine-containing beverages.
17. Participation in any other clinical drug study within 3 months before the IMP administration of this study.
18. Donation of blood within 3 months before the IMP administration.
19. Any medical or surgical procedure planned during the study period.
20. Male subjects who are sexually active with a female partner of childbearing potential and do not agree to use two medically accepted methods of contraception during the study and for three months after the dosing, and refrain from donating sperm during this time.
21. Female subjects for Part 2 need to be postmenopausal for at least one (1) year before participation or be surgically sterilized.
22. For subjects in Part 2, any indication of increased intracerebral pressure by neurological examination at inclusion, or another contraindication for LP.
23. Large tattoo or another condition of the skin or subcutaneous tissue that would prevent reliable assessment of local IREs.
24. Significant risk of suicidal behaviour, defined using the C-SSRS.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 8 +/- 1 days
  Incidence, type and severity of treatment-emergent AEs
Physical examination | 8 +/- 1 days
  Incidence of clinically significant physical examination findings
Vital signs | 8 +/- 1 days
  Incidence of clinically significant findings in systolic and diastolic blood pressure, heart rate and body temperature
12-lead electrocardiogram (ECG) | 24 hours
  Incidence of clinically significant findings in heart rate, PR interval, RR, QRS interval and QTcF
Pulse oximetry | 8 hours
  Incidence of clinically significant changes in blood oxygen saturation
Laboratory safety assessments - Haematology | 8 +/- 1 days
  Incidence of clinically significant laboratory variables in haemoglobin, erythrocytes, leucocytes, thrombocytes, mean corpuscular volume (MCV), mean corpuscular haemoglobin concentration (MCHC) and differential leucocyte count
Laboratory safety assessments - Clinical chemistry | 8 +/- 1 days
  Incidence of clinically significant laboratory variables in alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT), bilirubin total, bilirubin conjugated, albumin, creatinine, glucose, sodium, potassium, calcium, C-reactive protein (CRP), creatine kinase (CK), thyroid-stimulating hormone (TSH) and prolactin
Laboratory safety assessments - Coagulation | 8 +/- 1 days
  Incidence of clinically significant laboratory variables in plasma activated partial thromboplastin time (P-APTT) and international normalized ratio (INR)
Laboratory safety assessments - Urinalysis | 8 +/- 1 days
  Incidence of clinically significant laboratory variables in pH, erythrocytes, leukocytes, nitrite, protein, glucose and ketones
Laboratory safety assessments - CSF (Part 2 only) | 12 hours
  Incidence of clinically significant laboratory variables in cell count and protein concentration
Columbia-Suicide Severity Rating Scale (C-SSRS) | 8 +/- 1 days
  Incidence of subjects with increased suicidal tendencies measured by C-SSRS questionnaire consisting of maximum of 4 sections.
  Suicidal ideation: 5 yes/no questions with "yes" indicating suicidal ideation and "no" indicating no suicidal ideation.
  Intensity of ideation: 5 questions to be rated with respect to the most severe type if ideation (5 being the most severe intensity and 1 being the least intensity).
  Suicidal behavior: 5 yes/no questions with "yes" indicating suicidal behavior and "no" indicating no suicidal behavior.
  Actual attempts only: 2 questions to be rated with respect to the most severe outcome of the suicide attempt (highest score indicating the most severe outcome and 0 indicating no harm).

SECONDARY OUTCOMES:
HER-096 concentration levels | 24 hours
  Changes in HER-096 concentration levels in plasma and urine
HER-096 concentration in CSF (Part 2 only) | 12 hours
  Changes in HER-096 concentration levels in CSF

CONTACTS AND LOCATIONS:
Overall Officials: Aleksi Tornio, MD, Principal Investigator — Clinical Research Services Turku - CRST Oy
Locations (1):
- Clinical Research Services Turku - CRST Oy, Turku, Finland